CLINICAL TRIAL: NCT02564783
Title: The Burden of Pediatric Surgical Conditions in Rural Kenya - a Prospective Cohort Study
Brief Title: The Burden of Pediatric Surgical Conditions in Rural Kenya
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Veikko Schepel, Resident, Department of Plastic Surgery, Helsinki University Central Hospital
Other Study IDs: VSKENDU-1
Record Dates: First submitted 2015-09-22; First posted 2015-10-01 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Burden of Surgical Disease in Western Kenya

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
PURPOSE OF THE STUDY

The main purpose of this study is to find out what is the true burden of surgical conditions in pediatric population in a well defined geographical rural area in western Kenya.

DETAILED DESCRIPTION:
MATERIAL This research will be conducted in the Homa Bay county in western Kenya in previously selected locations around the county in rural area. An estimated 800 children and youth under the age of 18 will be selected for this study. This study will take place between October and November 2015. The investigators hypothesis, based on prior survey studies done in Sub-Saharan Africa, is that roughly 6% of the people under 18 are suffering from a surgical condition. In a sample size of 800 people the margin of error is 1,65%.

People who are currently being treated in a hospital will be excluded from the study. Also the people who decline from the study will be excluded. The number of declinations will be recorded.

METHODS The people will receive a written and a verbal information regarding the study and its purposes from the primary research assistant. If they decide to participate in the study they or their parent/guardian will be asked to sign an informed consent. Local interpreter will be available to help with possible questions.

The primary research assistant will conduct a short interview. Prior medical history will be taken. The participants will be asked their age. If age is not known the primary research assistant will estimate it. The height, weight and sex will be registered. A full physical examination will then be conducted. In this examination the participants will be assessed for visible deformations i.e. masses, scars, limb deformities. It will be determined whether the deformation is congenital or acquired. If the deformity is acquired the cause will be asked from the subject. The range of major joints will be registered. In case of palpable masses the possible diagnosis will be figured out using basic clinical skills. A structured survey sheet will be used collect the information. No other forms of diagnostic measures will be used. No blood or microbial culture samples will be collected and no x-ray imaging will be done.

If a surgical condition is diagnosed the participant will be informed about the nature and possible cause of this condition. No treatment procedures will be done on site.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18

Exclusion Criteria:

* Not meeting the age criteria.
* Declining to participate in the study.
* Patients who meet the criteria but are currently being treated in a hospital.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 800 children and youth under the age of 18 in a well defined area in rural Western Kenya (Kabondo city in Homa Bay County).
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of surgical conditions in population under 18 in rural Western Kenya | 25days (October 5th - October 30th 2015)

CONTACTS AND LOCATIONS:
Overall Officials: Erkki Tukiainen, Professor, Study Director — Helsinki University Hospital, Department of Plastic Surgery
Locations (1):
- Homa Bay County School District, Homa Bay County, Kenya